CLINICAL TRIAL: NCT02337712
Title: Once-daily Simultaneous Modulated Accelerated Thoracic Radiotherapy Compared With Twice-daily Radiotherapy in Limited Small-cell Lung Cancer Treated Concurrently With Cisplatin and Etoposide
Brief Title: Once-daily Simultaneous Modulated Accelerated Thoracic Radiotherapy in Limited Small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hui Liu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-FXY-037
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Small Cell Lung Cancer
Keywords: Small cell lung cancer; Radiotherapy; Dose fractionation
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- q.d. RT (Experimental): q.d. RT (65 Gy in 26 fractions) to the chest and concurrent etoposide and cisplatin
  Interventions: Radiation: q.d. RT; Drug: etoposide and cisplatin
- b.i.d.RT (Active Comparator): b.i.d.RT (45Gy in 30 fractions) to the chest and concurrent etoposide and cisplatin
  Interventions: Radiation: b.i.d.RT; Drug: etoposide and cisplatin

INTERVENTIONS:
Radiation: q.d. RT — 65 Gy in 26 fractions
  Arms: q.d. RT
Radiation: b.i.d.RT — 45 Gy in 30 fractions
  Arms: b.i.d.RT
Drug: etoposide and cisplatin — etoposide and cisplatin concurrent with radiotherapy

SUMMARY:
This Phase II randomized study is to determine whether once-daily simultaneous modulated accelerated thoracic radiotherapy (RT) resulted in better survival than twice-daily RT for patients with limited-stage small-cell lung cancer (LD-SCLC).

DETAILED DESCRIPTION:
This Phase II randomized study is to determine whether once-daily (qd)simultaneous modulated accelerated thoracic radiotherapy resulted in better survival than twice-daily(bid) RT for patients with limited-stage small-cell lung cancer (LD-SCLC).

All patients receive four to six cycles of etoposide and cisplatin (EP) every 3 weeks. Thoracic RT is initiated with cycle 1-3 of chemotherapy. Qd RT includes the delivery of 65 Gy in 26 fractions delivered on weekdays for a total of 33 days. Bid RT includes the delivery of 45 Gy in 30 fractions delivered on weekdays for a total of 19 days. After the chest RT and the last cycle of EP, prophylactic cranial irradiation is administered to those patients with a complete or partial remission.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of SCLC. Imaging studies' confirmation of limited stage.
* No previous chest radiotherapy, chemotherapy or biotherapy.
* Patients have measurable or evaluable lesions based on the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* White blood cell count ≥4×109 /L, platelet count≥100×109 /L, hemoglobin ≥100 g /L; serum creatinine and total bilirubin 1.5 times or less the upper limits of normal (ULN), aspartate aminotransferase two times or less the ULN.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Weight loss ≤10% within the past 3 months.
* Forced expiratory volume in 1 s >1 L.

Exclusion Criteria:

* Previous or recent another malignancy.
* A myocardial infarction within 6 months or had uncontrolled congestive heart failure, uncontrolled arrhythmia.
* Malignant pleural or pericardial effusion.
* Pregnant or Lactating.
* Weight loss >10% within the past 3 months.
* Drug addiction, long-term alcohol abuse and AIDS patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-01; Primary Completion 2020-09-30 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hui Liu, Professor, Principal Investigator — Sun yat-sen universtiy cancer center
Locations (1):
- Sun yat-sen university cancer center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Kong FM, Lally BE, Chang JY, Chetty IJ, Decker RH, Ginsburg ME, Kestin LL, Langer CJ, Movsas B, Videtic GM, Willers H, Rosenzweig KE; Expert Panel on Radiation Oncology-Lung. ACR Appropriateness Criteria(R) radiation therapy for small-cell lung cancer. Am J Clin Oncol. 2013 Apr;36(2):206-13. doi: 10.1097/COC.0b013e31827e5523. PMID 23511336
- [Background] Socinski MA, Bogart JA. Limited-stage small-cell lung cancer: the current status of combined-modality therapy. J Clin Oncol. 2007 Sep 10;25(26):4137-45. doi: 10.1200/JCO.2007.11.5303. PMID 17827464
- [Background] Turrisi AT 3rd, Kim K, Blum R, Sause WT, Livingston RB, Komaki R, Wagner H, Aisner S, Johnson DH. Twice-daily compared with once-daily thoracic radiotherapy in limited small-cell lung cancer treated concurrently with cisplatin and etoposide. N Engl J Med. 1999 Jan 28;340(4):265-71. doi: 10.1056/NEJM199901283400403. PMID 9920950
- [Background] Chen GY, Jiang GL, Wang LJ, Qian H, Fu XL, Yang H, Wu KL, Zhao S. Cisplatin/etoposide chemotherapy combined with twice daily thoracic radiotherapy for limited small-cell lung cancer: a clinical phase II trial. Int J Radiat Oncol Biol Phys. 2005 Jan 1;61(1):70-5. doi: 10.1016/j.ijrobp.2004.04.058. PMID 15629596
- [Background] Hu X, Bao Y, Zhang L, Guo Y, Chen YY, Li KX, Wang WH, Liu Y, He H, Chen M. Omitting elective nodal irradiation and irradiating postinduction versus preinduction chemotherapy tumor extent for limited-stage small cell lung cancer: interim analysis of a prospective randomized noninferiority trial. Cancer. 2012 Jan 1;118(1):278-87. doi: 10.1002/cncr.26119. Epub 2011 May 19. PMID 21598237
- [Background] Choi NC, Herndon JE 2nd, Rosenman J, Carey RW, Chung CT, Bernard S, Leone L, Seagren S, Green M. Phase I study to determine the maximum-tolerated dose of radiation in standard daily and hyperfractionated-accelerated twice-daily radiation schedules with concurrent chemotherapy for limited-stage small-cell lung cancer. J Clin Oncol. 1998 Nov;16(11):3528-36. doi: 10.1200/JCO.1998.16.11.3528. PMID 9817271
- [Background] Roof KS, Fidias P, Lynch TJ, Ancukiewicz M, Choi NC. Radiation dose escalation in limited-stage small-cell lung cancer. Int J Radiat Oncol Biol Phys. 2003 Nov 1;57(3):701-8. doi: 10.1016/s0360-3016(03)00715-6. PMID 14529774
- [Background] Miller AA, Wang XF, Bogart JA, Hodgson LD, Rocha Lima CM, Radford JE, Vokes EE, Green MR; Cancer and Leukemia Group B (CALGB). Phase II trial of paclitaxel-topotecan-etoposide followed by consolidation chemoradiotherapy for limited-stage small cell lung cancer: CALGB 30002. J Thorac Oncol. 2007 Jul;2(7):645-51. doi: 10.1097/JTO.0b013e318074bbf5. PMID 17607121
- [Background] Bogart JA, Herndon JE 2nd, Lyss AP, Watson D, Miller AA, Lee ME, Turrisi AT, Green MR; Cancer and Leukemia Group B study 39808. 70 Gy thoracic radiotherapy is feasible concurrent with chemotherapy for limited-stage small-cell lung cancer: analysis of Cancer and Leukemia Group B study 39808. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):460-8. doi: 10.1016/j.ijrobp.2003.10.021. PMID 15145163
- [Background] Liao ZX, Komaki RR, Thames HD Jr, Liu HH, Tucker SL, Mohan R, Martel MK, Wei X, Yang K, Kim ES, Blumenschein G, Hong WK, Cox JD. Influence of technologic advances on outcomes in patients with unresectable, locally advanced non-small-cell lung cancer receiving concomitant chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3):775-81. doi: 10.1016/j.ijrobp.2009.02.032. Epub 2009 Jun 8. PMID 19515503
- [Background] Shirvani SM, Juloori A, Allen PK, Komaki R, Liao Z, Gomez D, O'Reilly M, Welsh J, Papadimitrakopoulou V, Cox JD, Chang JY. Comparison of 2 common radiation therapy techniques for definitive treatment of small cell lung cancer. Int J Radiat Oncol Biol Phys. 2013 Sep 1;87(1):139-47. doi: 10.1016/j.ijrobp.2013.05.040. PMID 23920393
- [Background] Xia B, Chen GY, Cai XW, Zhao JD, Yang HJ, Fan M, Zhao KL, Fu XL. Is involved-field radiotherapy based on CT safe for patients with limited-stage small-cell lung cancer? Radiother Oncol. 2012 Feb;102(2):258-62. doi: 10.1016/j.radonc.2011.10.003. Epub 2011 Nov 5. PMID 22056536
- [Background] Murray N, Coy P, Pater JL, Hodson I, Arnold A, Zee BC, Payne D, Kostashuk EC, Evans WK, Dixon P, et al. Importance of timing for thoracic irradiation in the combined modality treatment of limited-stage small-cell lung cancer. The National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 1993 Feb;11(2):336-44. doi: 10.1200/JCO.1993.11.2.336. PMID 8381164
- [Background] Giuliani ME, Lindsay PE, Sun A, Bezjak A, Le LW, Brade A, Cho J, Leighl NB, Shepherd FA, Hope AJ. Locoregional failures following thoracic irradiation in patients with limited-stage small cell lung carcinoma. Radiother Oncol. 2012 Feb;102(2):263-7. doi: 10.1016/j.radonc.2011.12.009. Epub 2012 Jan 28. PMID 22285072
- [Background] Fan TY, Xing J, Lu J, Liu TH, Xu M, Zhang YJ, Shao Q, Li JB, Yu JM. Phase I/II study of induction chemotherapy plus concurrent chemotherapy and SMART-IMRT-based radiotherapy in locoregionally-advanced nasopharyngeal cancer. Oncol Lett. 2013 Mar;5(3):889-895. doi: 10.3892/ol.2013.1137. Epub 2013 Jan 15. PMID 23426016
- [Background] Yee D, Hanson J, Butts C, Reiman A, Joy A, Smylie M, Fenton D, Chu Q, Roa W. Phase I dose escalation trial of hypofractionated limited-field external beam thoracic radiotherapy for limited-stage small cell carcinoma of the lung. Radiother Oncol. 2010 Jul;96(1):78-83. doi: 10.1016/j.radonc.2010.05.013. Epub 2010 Jun 11. PMID 20542346
- [Derived] Qiu B, Li Q, Liu J, Huang Y, Pang Q, Zhu Z, Yang X, Wang B, Chen L, Fang J, Lin M, Jiang X, Guo S, Guo J, Wang D, Liu F, Chu C, Huang X, Xie C, Liu H. Moderately Hypofractionated Once-Daily Compared With Twice-Daily Thoracic Radiation Therapy Concurrently With Etoposide and Cisplatin in Limited-Stage Small Cell Lung Cancer: A Multicenter, Phase II, Randomized Trial. Int J Radiat Oncol Biol Phys. 2021 Oct 1;111(2):424-435. doi: 10.1016/j.ijrobp.2021.05.003. Epub 2021 May 13. PMID 33992717